CLINICAL TRIAL: NCT01422161
Title: Botulinum Toxin Type A Therapy as a Plasticity Inducing Agent for Recovery of Hand Function After Stroke
Brief Title: Study of Botulinum Toxin and Recovery of Hand Function After Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10-01126; 10-01126 (Other: Institutional Review Board (IRB) - NYU School of Medicine)
Record Dates: First submitted 2011-08-19; First posted 2011-08-23 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Stroke With Hemiparesis
Keywords: Rehabilitation; Fingers; Grasp; Hand; Strength; Brain Infraction; Pathology; Physiopathology; Functional Laterality; Neuronal Plasticity; Psychomotor Performance; Biomechanics; Touch; Weight-Bearing
MeSH Terms: interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum Toxin commonly known as BOTOX® (Experimental): Some subjects will receive BOTOX® injections. Subject will not be informed of what injection they received.
  Interventions: Drug: Botulinum Toxin commonly known as BOTOX®
- Placebo (Placebo Comparator): Some subject will receive a safe Placebo injection. Subjects will not be informed of what injection they have received.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin commonly known as BOTOX® — A total dose between 200-300 units of Botulinum toxin will be administered across 12 muscles of the affected hand.
  There will be 1 treatment cycle during the 9 week study.
  Other Names: BOTOX®; Saline
  Arms: Botulinum Toxin commonly known as BOTOX®
Drug: Placebo — The control group will receive a placebo injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether injections of botulinum toxin (commonly known as BOTOX®) into the affected hand of Stroke patients, while targeting the muscles controlling the hand, will lead to improved use of the hand when compared to injections of placebo (a substance that looks similar to the study drug but contains no active study medication).

DETAILED DESCRIPTION:
Hemiparesis is the most common motor impairment after stroke that frequently leads to persistent deficits in hand function. This study investigates whether the application of botulinum toxin to a set of synergistically-acting hand muscles, in conjunction with task-specific therapy, will lead to reorganization and improved motor function in the stroke-involved hand. The investigators will use objective psychophysical measures of hand function and hand function rating scales to investigate if Botox in conjunction with task-specific therapy will lead to:

* improved motor execution,
* improved motor planning during a psychophysical two-finger grasping and lifting task with varying object weight, and
* increased hand function as assessed by the time taken to complete fine motor tasks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to follow study instructions and likely to complete all required visits
* Ability to comply with the therapy protocol as assessed by the investigator
* 3 months post first-time unilateral stroke with right or left hemiparesis and complaints of unilateral hand dysfunction
* Must have ability to grasp and lift the test object
* Subjects must have upper extremity motor impairment

Exclusion Criteria:

* Known allergy or sensitivity to botulinum toxin type A (BOTOX).
* Females with a positive pregnancy test, or who are breast-feeding, planning a pregnancy during the study, who think that they may be pregnant at the start of the study or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
* Concurrent participation in another investigational drug or device study or participation in another Botulinum toxin study in the 6 months prior to study.
* Treatment with botulinum toxin of any serotype in the 3 months prior to study enrollment
* Any medical condition that may put the subject at increased risk with exposure to BOTOX including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amytrophic lateral sclerosis, or any other disorder that might interfere with neuromuscular function.
* Evidence of alcohol, drug abuse or other relevant neuropsychiatric condition.
* Infection or skin disorder at an anticipated injection site.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* History of surgery or other significant injury to either upper extremity causing mechanical limitations that preclude task performance.
* Previous neurological illness such as head trauma, prior stroke, epilepsy, or demyelinating disease.
* Complicating medical problems such as uncontrolled hypertension, diabetes with signs of polyneuropathy, severe renal, cardiac or pulmonary disease, or evidence of other concurrent neurologic or orthopedic conditions precluding the subject from complying with the study protocol.
* Current treatment with intrathecal baclofen.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Raghavan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sample size is estimated based on a treatment difference of 20% between the two groups
Groups:
- Botulinum Toxin Commonly Known as BOTOX®: Some subjects will receive BOTOX® injections. Subject will not be informed of what injection they received.
  Botulinum Toxin commonly known as BOTOX®: A total dose between 200-300 units of Botulinum toxin will be administered across 12 muscles of the affected hand.
Period: Overall Study
Arm/Group | Botulinum Toxin Commonly Known as BOTOX® | Placebo
Started | 10 | 6
Completed | 10 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Botulinum Toxin Commonly Known as BOTOX®: Some subjects will receive BOTOX® injections. Subject will not be informed of what injection they received.
  Botulinum Toxin commonly known as BOTOX®: A total dose between 200-300 units of Botulinum toxin will be administered across 12 muscles of the affected hand.
  The control group will receive a placebo injection. There will be 1 treatment cycle during the 9 week study.
- Placebo: Some subject will receive a safe Placebo injection. Subjects will not be informed of what injection they have received.
  Botulinum Toxin commonly known as BOTOX®: A total dose between 200-300 units of Botulinum toxin will be administered across 12 muscles of the affected hand.
  The control group will receive a placebo injection. There will be 1 treatment cycle during the 9 week study.
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Commonly Known as BOTOX® | Placebo | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Time Taken to Form a Stable Grasp Pre-Treatment
Description: Assessments are done on day 1, before the 1st Botulinum toxin injection.
  They will be assessed for:
  * Hand motor impairment (execution and planning) during a functional grasp and lift tasks.
  * Hand function.
Time Frame: Day 1
Population: Improved motor execution as measured by the time taken to form a stable grasp.
Measure: Mean (Standard Error); unit: Preload phase duration in Seconds
Groups:
- Control (Saline) Group -PRE Treatment: Some subjects will receive BOTOX® injections. Subject will not be informed of what injection they received.
  Botulinum Toxin commonly known as BOTOX®: A total dose between 200-300 units of Botulinum toxin will be administered across 12 muscles of the affected hand.
  The control group will receive a placebo injection. There will be 1 treatment cycle during the 9 week study.
- Botox Group -PRE Treatment: A total dose between 200-300 units of Botulinum toxin will be administered across 12 muscles of the affected hand.
  There will be 1 treatment cycle during the 9 week study.
Arm/Group | Control (Saline) Group -PRE Treatment | Botox Group -PRE Treatment
Number analyzed (Participants) | 6 | 10
Preload phase duration in Seconds | 1.51 (.21) | 1.14 (.59)

2. Primary Outcome: Time Taken to Form a Stable Grasp Post Treatment
Description: * Hand motor impairment (execution and planning) during a functional grasp and lift tasks.
  * Hand function.
Time Frame: 90 Days
Population: Time taken to form a stable grasp.
Measure: Mean (Standard Error); unit: Preload phase duration in Seconds
Groups:
- Control (Saline) Group -POST Treatment: Some subject will receive a safe Placebo injection. Subjects will not be informed of what injection they have received.
  Botulinum Toxin commonly known as BOTOX®: A total dose between 200-300 units of Botulinum toxin will be administered across 12 muscles of the affected hand.
  The control group will receive a placebo injection. There will be 1 treatment cycle during the 9 week study.
- Botox Group -POST Treatment: A total dose between 200-300 units of Botulinum toxin will be administered across 12 muscles of the affected hand.There will be 1 treatment cycle during the 9 week study.
Arm/Group | Control (Saline) Group -POST Treatment | Botox Group -POST Treatment
Number analyzed (Participants) | 6 | 10
Preload phase duration in Seconds | 2.65 (0.17) | .79 (.09)

3. Secondary Outcome: Measure of Upper Limb Motor Impairment Measured by Fugl Meyer Scale
Description: This scale has 3 points for each item. A zero is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. Reflex activity is measured using 2 points only, with a score of 0 or 3 for absence and presence of reflex. The maximum total score that can be obtained in Fugl Meyer assessment is 226, though it is common practice to assess all domains separately.The five domains assessed by Fugl-Meyer scale are:
  Motor function (Maximum score in upper limb = 66; Maximum score in lower limb = 34) Sensory function (Maximum score = 24) Balance (Maximum score = 14) Range of motion of joints (Maximum score = 44) Joint pain (Maximum score = 44)
Time Frame: Pre-Treatment, Day 90
Population: Total upper limb Fugl Meyer scale score out of 66.
Measure: Mean (Standard Error); unit: Fugl Meyer Scale Score
Arm/Group | Control (Saline) Group -PRE Treatment | Botox Group -PRE Treatment
Number analyzed (Participants) | 6 | 10
Fugl Meyer Scale Score | 47.6 (4) | 40.7 (3.31)

4. Secondary Outcome: Disability Measured by Modified Rankin Scale Score Post-Treatment
Description: Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.The mRS is an ordered scale coded from 0 (no symptoms at all), 1 (No significant disability despite symptoms; able to carry out all usual duties and activities), 2 (Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance), 3 (Moderate disability; requiring some help, but able to walk without assistance), 4 (Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance), 5 (severe disability) and 6 (death).
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: Modified Rankin Scale Score
Arm/Group | Control (Saline) Group -POST | Botox Group -POST
Number analyzed (Participants) | 6 | 10
Modified Rankin Scale Score | 2 (0.36) | 1.8 (0.24)

5. Secondary Outcome: Motor Impairment Measured by the Fugl-Meyer Scale Post-Treatment
Description: Scale is comprised of five domains and there are 155 items in total: Motor functioning (in the upper and lower extremities); Sensory functioning (evaluates light touch on two surfaces of the arm and leg, and position sense for 8 joints); Balance (contains 7 tests, 3 seated and 4 standing); Joint range of motion (8 joints); Joint pain. Each domain contains multiple items, each scored on a 3-point ordinal scale (0 = cannot perform, 1= perform partially, 2 = perform fully).
Time Frame: 1 Day and 90 Days
Population: Total upper limb Fugl Meyer Score out of 66.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control (Saline) Group -POST Treatment | Botox Group -POST Treatment
Number analyzed (Participants) | 6 | 10
score on a scale | 52.1 (3.5) | 45.5 (2.85)

6. Secondary Outcome: Disability Measured by Modified Rankin Scale Score Pre-Treatment
Description: as for outcome 4
Time Frame: Pre-Treatment
Measure: Mean (Standard Deviation); unit: Modified Rankin Scale Score
Arm/Group | Control (Saline) Group -Pre | Botox Group -Pre
Number analyzed (Participants) | 6 | 10
Modified Rankin Scale Score | 2.3 (.33) | 2.6 (.33)

ADVERSE EVENTS:
Time Frame: 90 Days
Arm/Group | Botulinum Toxin Commonly Known as BOTOX® | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes